CLINICAL TRIAL: NCT01859234
Title: Evaluation of VEGF Expression With 89Zr-bevacizumab PET Scan in Patients With Relapsing Multiple Myeloma; a Feasibility Study
Brief Title: 89Zr-bevacizumab PET Scan in Patients With Relapsing Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, E.G.M. de Waal, Hematologist, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCGABR40641
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; PET scan
MeSH Terms: conditions — Multiple Myeloma | interventions — 89Zr-bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 89Zr-bevacizumab PET scan (Experimental): all patients included in the study will have a 89Zr-bevacizumab PET scan
  Interventions: Drug: 89Zr-bevacizumab

INTERVENTIONS:
Drug: 89Zr-bevacizumab — 89Zr-bevacizumab will only be given once, prior for the PET scan. 5 mg will be given iv.
  Other Names: Bevacizumab Roche registration limited eu/1/04/300/001; 89Zr-bevacizumab ATC code L01XC07

SUMMARY:
The purpose of this study is to see whether 89Zr-bevacizumab PET scanning is feasible in relapsing multiple myeloma patients.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a clonal B cell disorder characterised by a monoclonal plasma cell population in bone marrow, with bone pain, anaemia, hypercalcaemia, and kidney dysfunction as clinically presenting symptoms. Osseous involvement is one of the most predominant features of patients with MM; 90% of the patients develop lytic bone lesions. Lytic bone lesions are the result of increased bone resorption and reduced bone formation. The regular method to detect bone lesions is skeletal survey. This technique can only detect lesions that have lost 30% or more of the trabecular bone. Another weakness is the fact that lesions persist after treatment with chemotherapy or radiotherapy and no clear distinction can be made whether vital tumour cells persist in these lesions. New bone lesions are a sign of disease progression. Furthermore they give clinical signs as bone pain and in the worse case scenario pathological fractures. Alternative scanning methods have been developed to visualize the malignant plasma for example by making use of enhanced metabolic activity of the plasma cells defined by the uptake of 18F-fluorodeoxyglucose -Positron Emission tomography (FDG-PET. The use of FDG-PET in newly diagnosed MM patients is well studied.

The increased FDG-uptake by the tumour is related to a high metabolic activity. This might be a consequence of tumour hypoxia causing new vessel formation. There seems to be a relationship between MM and angiogenesis, the formation of new blood vessels from exciting blood vessels. There is an increased microvessel density (MVD) of the affected bone marrow in patients with active MM. Vascular endothelial growth factor (VEGF) is an important mediator of angiogenesis. MM cell lines were found to express VEGF mRNA and secrete the protein in the extracellular environment thereby stimulating angiogenesis.

Inhibition of the process of angiogenesis is used in the treatment of MM, for instance by means of thalidomide and lenalidomide. Blocking VEGF itself can be obtained by means of bevacizumab, a recombinant, humanised monoclonal antibody that binds to all isoforms of human VEGF with high affinity. Treatment with bevacizumab is well established in solid tumours, like colon cancers and renal cell carcinomas and is currently tested in acute myeloid leukaemia and MM.

VEGF imaging with radiolabeled bevacizumab has been developed. Bevacizumab binds VEGF and can be labeled with the PET isotope Zirconium-89 (89Zr) while preserving VEGF binding properties. In a human ovarian tumor xenograft, PET imaging 24 hours after injection of 89Zr-bevacizumab showed high uptake in well perfused organs and in the tumor.

The high VEGF production by myeloma cells makes VEGF a very interesting target for tumor visualization. 89Zr-bevacizumab PET imaging could be more sensitive for myeloma lesions.

So, in conclusion, VEGF is expressed by MM plasma cells, thereby providing a rationale that the assessment of VEGF-levels in the micro-environment of MM tumors could potentially be used as a diagnostic tool to see if there is disease activity. Especially in the relapsed setting this is of invaluable importance, since conventional skeletal survey has limitations in this setting. Furthermore, 89Zr-bevacizumab PET imaging could provide information about treatment options and treatment response.

ELIGIBILITY:
Inclusion Criteria:

Patients with relapsing multiple myeloma according to international defined guidelines:

Relapse after having achieved complete remission:

1. Reappearance of paraprotein
2. More than 5% plasma cells in bone marrow.
3. New lytic lesions or progression of old lesions.
4. New hypercalcaeamia.

Relapse after having achieved partial remission

1. Increases of paraprotein with more than 25%
2. Increase of urine paraprotein with more than 25%
3. Increase of plasma cells in bone marrow with 10%
4. New lytic lesions or progression of old lesions
5. New hypercalcaemia -

Exclusion Criteria:

Radiotherapy in the last 3 months.

* Ineligible to lay supine during the PET scan.
* Age ≤18 years.
* Pregnancy.
* Claustrophobia
* Severe kidney dysfunction; serum-creatinine ≥250 µM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Focal lesion of 89Zr-bevacizumab PET scanning in patients with relapsing multiple myeloma | during scanning
  We assume focal lesion will be feasible with 89Zr-bevacizumab PET scanning in patients with relapsing multiple myeloma. For each 89Zr-bevacizumab PET scan the amount of focal lesion and the localisation will be reported. When there is diffuse bone marrow uptake this will also be reported. The focal lesion found on the 89Zr-bevacizumab PET scan will be compared with focal lesions found on the FDG-PET scan. Furthermore the amount of focal lesion will be compared with the expression of VEGF, MVD, HIF 1 alpha and 2 alpha and GLUT 1 and 3.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands